CLINICAL TRIAL: NCT00258635
Title: A Double-Blind Phase IIb Study to Evaluate the Safety and Efficacy of Different Doses of Tyrosine Adsorbed Ragweed Allergoid With MPL® With a Single-Blind Portion to Evaluate the Residual Allergenicity in Skin Test in Patients Sensitized to Ragweed Pollen.
Brief Title: Investigation of Safety+Efficacy of Different Doses of RagweedMATAMPL;Assessment of Residual Allergenicity Using Skin Prick Test
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RagweedMATAMPL203
Record Dates: First submitted 2005-11-25; First posted 2005-11-28 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Specific Immunotherapy
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Biological: RagweedMATAMPL

SUMMARY:
The purpose of this study is to assess the immunological differences between three RagweedMATAMPL treatment arms compared to placebo with respect to immunoglobulin levels.

In addition, the study will assess the reduced allergenicity of modified Ragweed Pollen contained in RagweedMATAMPL compared to unmodified native allergen using skin prick testing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be male or female aged 18-50 years, inclusive.
2. Patients must have a positive skin prick test for ragweed allergen (wheal that is ≥5 mm larger than the negative control).
3. Positive skin prick test to positive histamine control with a wheal (longest) diameter ≥3 mm.
4. Negative skin prick test to negative control (redness, but no wheal is acceptable).
5. Specific IgE for ragweed as documented by radioallergosorbent or equivalent test with class ≥2.
6. History of at least 1 season of moderate to severe seasonal rhinoconjunctivitis due to an IgE - mediated allergy to pollen from ragweed as derived from the allergic history.
7. Patients must score in the disease severity questionnaire as moderate or severe.
8. Males or non-pregnant, non-lactating females who are post-menopausal or naturally or surgically sterile (hysterectomy; bilateral oophorectomy; bilateral tubal ligation with surgery at least 6 weeks prior to study initiation).

   Females of childbearing potential have a confirmed absence of pregnancy according to a negative urine pregnancy test and must be using one of the following acceptable birth control methods:
   1. Intrauterine device in place for at least 90 days;
   2. Barrier method (condom or diaphragm) with spermicide;
   3. Stable hormonal contraceptive for at least 90 days prior to study and through study completion;
   4. Abstinence;
   5. Non-heterosexual lifestyle;
   6. Vasectomized partner for at least 90 days.
9. Patients who are normally active and otherwise judged to be in good health on the basis of medical history, physical examination, and routine laboratory tests.
10. Patients must be willing and able to attend required study visits.
11. Patients must be able to follow instructions.
12. Patients must be willing and able to give written informed consent for this study. Consent must be obtained prior to initiation of any washout period.
13. Spirometry at Screening demonstrates FEV1 ≥ 80% predicted and FEV1/FVC ≥70%, when applicable

Exclusion Criteria:

1. Acute or subacute atopic dermatitis and/or urticaria factitia and/or urticaria due to physical or chemical influence and/or chronic dermatitis.
2. Patient has moderate to severe asthma.
3. Visual inspection of the forearms indicates potential problems with the conduct or interpretation of the skin prick test; both forearms must be available for testing.
4. History or presence of diabetes (insulin dependent and non-dependent), cancer or any clinically significant cardiac, metabolic renal, hematologic diseases or disorders.
5. Recent clinically significant history (within 2 years) of hepatic gastrointestinal, dermatologic, venereal, neurologic or psychiatric diseases or disorders.
6. Any clinically significant (as determined by the Investigator) abnormal laboratory value at Visit 1.
7. Clinically relevant sensitivity against perennial allergens [house dust mites (Dermatophagoides pteronyssinus, Dermatophagoides farinae), molds (Cladosporium cladosporioides, Alternaria alternata, Penicillium chrysogenum, Aspergillus fumigatus), cat epithelia (Felis domesticus), dog epithelia (Canis familiaris) and horse epithelia (Equus caballus)], documented by a positive case history, prick test wheal size ≥3 mm in diameter larger than the negative control or radioallergosorbent test with class ≥2. Exceptions: The Investigator may judge the sensitivity as not clinically relevant.
8. Clinically relevant sensitivity against seasonal allergens [mountain cedar, ash, birch, elm, maple, hickory, oak, cottonwood, bermuda grass and grass mix] documented by a positive case history, prick test wheal size ≥3 mm in diameter larger than the negative control or radioallergosorbent test with class ≥2. Exceptions: some or all of the listed allergens must not be tested if they are not common to the Investigator´s region or, if common to the region, no overlap exists between the allergen(s) season and the treatment and post treatment phase of the study. Furthermore, subjects will not be excluded if the Investigator may judge the sensitivity as not clinically relevant.
9. Secondary alteration at the affected organ (i.e. emphysema, bronchiectasis).
10. History of autoimmune diseases (e.g. of liver, kidney, thyroid, nervous system), and/or rheumatoid diseases.
11. Patient is taking ß-blockers for any indication including eye drops.
12. Patient who is not allowed to receive adrenalin.
13. Patients in whom tyrosine metabolism is disturbed, especially in the case of tyrosinemia and alkaptonuria.
14. Presence of a disease with a pathogenesis interfering with the immune response and patient has received medication which could influence the results of this study.
15. Documented evidence of acute or significant chronic infection.
16. History of anaphylaxis, including anaphylactic food allergy, insect venom anaphylaxis, exercise or drug induced anaphylaxis.
17. Documented history of angioedema.
18. Hypersensitivity to excipients in the study medications.
19. Previous or current immunotherapy with comparable ragweed allergen extracts.
20. Currently using anti-allergy medication and other drugs with antihistaminic activity.
21. Patients currently participating in a clinical trial or who have been exposed to study medication within the last 30 days.
22. Patients who cannot communicate reliably with the Investigator or who are not likely to cooperate with the requirements of the study.
23. Patient is pregnant or planning pregnancy and/or lactating.
24. Patient has received treatment with preparation containing MPL® during the past 12 months.
25. Concurrent use of any prohibited medication(s),or inadequate washout of any medication.
26. Any systemic disorder that could interfere with the evaluation of the study medication(s).
27. Clinical history (within 2 years) of drug or alcohol abuse that would, in the opinion of the Investigator, interfere with the patient's participation in the study.
28. Patient who has a positive urine drug screen (cocaine metabolites, cannabinoids, opiates, PCP, or amphetamine), or a positive alcohol saliva test.
29. Study site staff or immediate relatives of study site staff or other individuals who would have access to the clinical study protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2005-11; Primary Completion 2006-08-07 (Actual); Study Completion 2006-08-07 (Actual)

PRIMARY OUTCOMES:
To assess immunological differences between three Ragweed MATA MPL treatment arms compared to placebo with respect to immunoglobulin levels (ragweed spec. IgG, IgG1, IgG4,IgE). | 9 weeks

SECONDARY OUTCOMES:
Residual allergenicity of modified Ragweed pollen in RagweedMATAMPL compared to unmodified native allergen using Skin Prick Test; | 20 minutes and 6 hours after skin prick test
Tolerability of native, modified allergens and tyrosine adsorbents with and without MPL® using Skin Prick Test; | 20 minutes and 6 hours after skin prick test
Tolerability of different subcutaneous doses; | 9 weeks
Tolerability of the cumulative subcutaneous doses; | 9 weeks
Clinical chemistry, hematology and urinalysis; | 9 weeks
Number of Adverse Events (AEs); | 9 weeks
Number of Adverse Reactions; | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl Jürgen Fischer von Weikersthal-Drachenberg, MD, Study Chair — Allergy Therapeutics
Locations (4):
- United States (4):
  - Michigan Respiratory Health and Research Institute, Novi, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Regional Allergy & Asthma Consultants, Asheville, North Carolina
  - Lovelace Scientific Resources, Austin, Texas